CLINICAL TRIAL: NCT06017830
Title: The Effectiveness of Physical Therapy on Sexual Function in Patients With Low Back Pain
Brief Title: The Effect of Physical Therapy on Sexual Function
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 pandemi limited the number of patients who was applied physical therapy
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Gunay ER, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 48670771-514
Record Dates: First submitted 2021-06-25; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Sexual Dysfunction; Low Back Pain
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with low back pain (Experimental)
  Interventions: Device: Physical treatment agents

INTERVENTIONS:
Device: Physical treatment agents — Physical treatment agents such as TENS (transcutaneous electric nerve stimulation), hot pack and ultrasound will be applied to patients with low back pain. Sexual function will be assessed before, just after and 3 months later physical therapy.

SUMMARY:
Sexual function in low back pain and after lumbar surgery has been evaluated in many studies In a few studies, sexual function problems after surgery have also been reported. In the literature, there is no study that investigates the effectiveness of physical therapy on sexual function in patients with low back pain. In this study, the effectiveness of physical therapy on sexual function in patients with low back pain will be evaluated.

DETAILED DESCRIPTION:
63 patients who had chronic low back pain who applied to City Hospital, Physical Medicine and Rehabilitation Department between January 2021 and January 2023 were enrolled in the study. Sexually active patients between the ages of 18 and 60, for whom physical therapy was planned for low-back pain related to lumbar pathologies, were included in the study. Informed consent was obtained from all patients. Exclusion criteria were defined as having contraindications for any physical therapy agents, having cardiovascular, neurological, psychiatric disease, or sexual disorders.

Short Form-12 (SF-12), Oswestry Disability Index (ODI), and Hospital Anxiety and Depression Scale (HAD) were recorded. International Index of Erectile Function (IIEF) and Female Sexual Function Index (FSFI) were utilized to evaluate sexual function

Fifteen sessions of physical therapy were planned for each patient. The physical therapy program included 15 minutes of conventional transcutaneous electrical nerve stimulation, 10 minutes of ultrasound, and 15 minutes of superficial heaters such as hot packs or infrarouge. All patients were evaluated the day before the first physical therapy session, the one-month and three-month after the last physical therapy session.

ELIGIBILITY:
Inclusion Criteria:

* low back pain due to lumbar pathologies
* being sexually active
* have no contraindications for physical therapy agents

Exclusion Criteria:

* known sexual function problems,
* known psychiatric disease and/or are taking antidepressant
* diabetes mellitus,
* cardiovascular disease
* neurological diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
change from sexual function scores at just after physical therapy and 3 months | Before, just after and 3 months later physical therapy
  Female Sexual Function Index for women and International Index of Erectile Function for men will be used. There is no cut-off values. Better scores mean better results

SECONDARY OUTCOMES:
change from disability scores at just after physical therapy and 3 months | Before, just after and 3 months later physical therapy
  Oswestry Disability Index will be used. min-max 0-100. better scores means worse results
change from quality of life at just after physical therapy and 3 months | Before, just after and 3 months later physical therapy
  Short Form-12 will be used. min-max 0-100. better score means better quality of life.
change from mood at just after physical therapy and 3 months | Before, just after and 3 months later physical therapy
  Hospital Anxiety and Depression Scale will be used. min-max 0-21. better score means better result.

CONTACTS AND LOCATIONS:
Overall Officials: Gunay ER, Principal Investigator — Prof Dr Cemil Taşçıoğlu Şehir Hastanesi
Locations (1):
- Prof Dr Cemil Taşçıoğlu Şehir Hastanesi, Istanbul, Turkey (Türkiye)